CLINICAL TRIAL: NCT02441400
Title: EndoStim Patient Registry-LES Stimulation System for the Treatment of GERD
Brief Title: EndoStim Patient Registry
Acronym: RESTORE
Status: Terminated | Type: Observational
Why Stopped: Company no longer operational
Sponsor: EndoStim Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS500
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: GERD
Keywords: GERD; LES Pressure; Electrical Stimulation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EndoStim LES Stimulation System implant.: Registry subjects whom have been implanted commercially with the EndoStim LES Stimulation System device.
  Interventions: Device: EndoStim LES Stimulation System

INTERVENTIONS:
Device: EndoStim LES Stimulation System

SUMMARY:
To provide a research tool enabling physicians to monitor long term clinical outcomes for patients undergoing gastroesophageal reflux disease (GERD) treatment with EndoStim LES Stimulation System.

DETAILED DESCRIPTION:
The EndoStim Patient Registry provides a framework for data collection on patients with GERD treated with the EndoStim LES Stimulation System. The primary objective is to provide a tool for participating physician investigators to collect and analyze outcomes data related to the use of the EndoStim LES Stimulation System.

This is a prospective, multi-center patient Registry. Sites may choose to also retrospectively enroll previously treated patients (after obtaining informed consent) and enter retrospective data into case report forms paper or on-line.

ELIGIBILITY:
Inclusion Criteria:

1. Subject meets therapy indications
2. Subject signs informed consent
3. Subject has a planned EndoStim LES Stimulation System implant (prospective) OR subject has already had EndoStim LES Stimulation System implant (retrospective)

Exclusion Criteria:

1. Subject meets therapy contraindications

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of GERD who are undergoing or have already undergone EndoStim LES stimulation system implantation.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-05; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 5 years post-implant
  Safety will be assessed by incidence and severity of adverse events through 5 years of follow-up

SECONDARY OUTCOMES:
Change in GERD-HRQL | Change in GERD-HRQL questionnaire score will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline GERD-HRQL
Comparison of pH values | The pH values of % 24-hour esophageal pH < 4.0, and the number of reflux events > 1 minute and > 5 minutes will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline in the following (while off PPI): % 24-hour esophageal pH<4.0, and number of reflux events >1 minute and > 5 minutes
Comparison of symptoms and quality of life | Symptoms will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline in symptoms (measured by patient diary) and in quality of life (measured by SF-12)
Change in antisecretory medication use | The use of antisecretory medication will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline in antisecretory medication use
Change in Structured GI Questionnaire responses (vs. baseline) | Symptoms will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline on Structured GI Questionnaire responses
Change in sleep related quality of life | Sleep related quality of life will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline in sleep related quality of life (measured by Pittsburgh Sleep Quality Index)
Change in work productivity impairment | Work productivity will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline in work productivity impairment (measured by Work Productivity and Activity Impairment Questionnaire)
Change in Reflux Disease Questionnaire (RDQ) scores | RDQ questionnaire score will be assessed at baseline, 3-6 months post implant, and then annually until 5 years
  Change from baseline in RDQ scores

CONTACTS AND LOCATIONS:
Overall Officials: Virender K Sharma, MD, Study Director — EndoStim Inc.; Joachim Labenz, MD, Principal Investigator — Diakonie Klinikum
Locations (30):
- Fundacion Favaloro, Buenos Aires, Argentina
- University Hospital Vienna, Vienna, Austria
- Aarhus University Hospital, Aarhus, Denmark
- Germany (23):
  - SANA Klinikum Lichtenberg, Berlin
  - Evangelisches Krankenhaus Castrop-Rauxel, Castrop-Rauxel
  - Heilig Geist-Krankenhaus Köln, Cologne
  - St. Marienstift Krankenhaus Friesoythe, Friesoythe
  - Hospital zum Heiligen Geist Fritzlar, Fritzlar
  - Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - Wolfartklinik Graefelfing, Gräfelfing
  - Martha Maria Krankenhaus Halle-Dölau, Halle
  - Asklepios Klinik Altona, Hamburg
  - KRH Klinikum Siloah Hannover Oststadt, Hanover
  - Evangelisches Krankenhaus Herne, Herne
  - Klinikum Konstanz, Konstanz
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum Memmingen, Memmingen
  - Klinikum Minden Johannes Wesling, Minden
  - Klinikum Muenchen Bogenhausen, München
  - Friedrich-Ebert-Krankenhaus Neumünster, Neumünster
  - Asklepios Schwalm-Eder Kliniken GmbH, Schwalmstadt
  - Jung Stilling - Siegen, Siegen
  - St. Marien-Krankenhaus Siegen, Siegen
  - Klinikum Stuttgart, Krankenhaus Bad Cannstatt, Stuttgart
  - Ev. Krankenhaus Wesel GmbH, Wesel
- Hospital San José, Monterrey, Mexico
- Maastricht University Medical Center, Maastricht, Netherlands
- United Kingdom (2):
  - Spire Leicester Hospital, Leicester
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez L, Rodriguez P, Neto MG, Ayala JC, Saba J, Berel D, Conklin J, Soffer E. Short-term electrical stimulation of the lower esophageal sphincter increases sphincter pressure in patients with gastroesophageal reflux disease. Neurogastroenterol Motil. 2012 May;24(5):446-50, e213. doi: 10.1111/j.1365-2982.2012.01878.x. Epub 2012 Jan 31. PMID 22292889
- [Background] Rodriguez L, Rodriguez P, Gomez B, Ayala JC, Saba J, Perez-Castilla A, Galvao Neto M, Crowell MD. Electrical stimulation therapy of the lower esophageal sphincter is successful in treating GERD: final results of open-label prospective trial. Surg Endosc. 2013 Apr;27(4):1083-92. doi: 10.1007/s00464-012-2561-4. Epub 2012 Oct 17. PMID 23073680
- See also: Registry sponsor's website — http://www.endostim.com